CLINICAL TRIAL: NCT00003759
Title: Intravesical Treatment of Superficial Bladder Cancer Characterized on the Basis of the Tumor Markers p53 and pRb
Brief Title: AD 32 With or Without BCG After Surgery in Treating Patients With Newly Diagnosed or Recurrent Superficial Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anthra Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066883; ANTHRA-A9701/ID97-038; MDA-ID-97038
Record Dates: First submitted 1999-11-01; First posted 2003-07-18 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2002-11

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; recurrent bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine; valrubicin

INTERVENTIONS:
Biological: BCG vaccine
Drug: valrubicin
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies such as BCG use different ways to stimulate the immune system and stop cancer cells from growing. It is not yet known whether AD 32 is more effective with or without BCG after surgery for superficial bladder cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of AD 32 with or without BCG after surgery in treating patients who have newly diagnosed or recurrent superficial bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of peri-operative intravesical AD 32 alone or supplemented with BCG in patients with newly diagnosed or recurrent superficial bladder cancer characterized as either high risk or low risk based on the tumor markers p53 and pRb.
* For low-risk patients, assess the efficacy of peri-operative AD 32 in preventing tumor recurrence.
* For high-risk patients, assess the efficacy of combined intravesical therapy with AD 32 administered within 8 hours after transurethral resection along with BCG in decreasing the incidence of tumor progression.
* Evaluate systemic exposure and urine recovery of AD 32 through pharmacokinetic analysis in a subset of patients.

OUTLINE: This is a randomized, open-label study.

All patients undergo complete transurethral resection to remove bladder tumors. AD 32 is administered by catheter into the bladder within 8 hours after surgery. Patients must hold the AD 32 in the bladder for 90 minutes.

After pathological and tumor marker analysis, patients are assigned to the low or high-risk group as defined by their p53 and pRb phenotype.

* Low risk: Patients with carcinoma in situ receive BCG by catheter into the bladder once weekly for 6 weeks beginning 7-21 days after treatment with AD 32. Patients assigned to the low-risk group who do not have carcinoma in situ receive no further treatment.
* High-risk: Patients also receive BCG once weekly for 6 weeks and then once weekly for 3 weeks at 3 months, 6 months, and then every 6 months for a total of 3 years after the first BCG treatment.

All patients undergo cystoscopy every 3 months for the first year and then every 6 months for the next 2 years.

PROJECTED ACCRUAL: Approximately 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed or recurrent (at least 2 occurrences within 12 months) Ta, multifocal Ta (at least 2 visible tumors), or stage T1 bladder cancer

  * No carcinoma in situ (Tis) only
  * No T2 or greater tumors
* No evidence of upper tract (ureter or renal pelvic) transitional cell carcinoma based on intravenous pyelogram performed within 4 months of the TURB

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,500/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or superficial transitional cell carcinoma of the bladder

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biological response modifiers

Chemotherapy:

* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-11; Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin P. Dinney, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States